CLINICAL TRIAL: NCT06650345
Title: Exploring the Impact of Supervised Treadmill Aerobic Exercise on Cognitive Function and Apoptotic-Related Biomarkers in Aging Individuals
Brief Title: Aerobic Exercise Effects on Cognitive Function in Aging Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sami Gabr, Clinical investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RRC-2013-015
Record Dates: First submitted 2024-10-07; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Function; Exercise Training
Keywords: Cognitive abilities ,Apoptosis, LOTCA,exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The participants were categorized into two groups, specifically the control group (consisting of 30 individuals) and the exercise group (also comprising 30 individuals), based on their participation in an exercise program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (No Intervention): non-exercised participants with daily life activities
- exercise group (Experimental): participants engaged in a 12-week exercise regimen structured thrice weekly.Each session's intensity was customized to match the individual's maximum and resting heart rates. The warm-up involved stretching and a 5 to 10-minute walk. In the core exercise phase, participants aimed to reach their predetermined training heart rate (THR max; between 60 to 70%) for 45-60 minutes through intervals on a treadmill, bike, or stair climber.The exercise protocol was designed to elicit physical exertion equivalent to 30-45% of their maximum oxygen consumption (VO2 max)
  Interventions: Other: supervised aerobic exercise

INTERVENTIONS:
Other: supervised aerobic exercise — In this training program, the participants exercised for 45-60 minutes through intervals on a treadmill, bike, or stair climber, three times a week for 12 weeks.
  Arms: exercise group

SUMMARY:
Positive effects are exerted by participating in moderate exercise training with physical activity which positively affects body health, including cognitive abilities, among older adults. Thus, the investigators are trying to study the potential effects of the supervised aerobic training regimen for 12 weeks on cognitive function among older adults based on molecular changes in cellular apoptosis.

DETAILED DESCRIPTION:
Physical activity exerts many positive effects on body health, including cognitive abilities, among older adults. Nevertheless, a paucity of knowledge exists regarding the potential anti-apoptotic benefits of moderate exercise and its potential influence on cognitive function. The objective of the present study was to explore the possible connection between the anti-apoptotic mechanisms associated with exercise and cognitive performance in a cohort of 60 older adults who participated in a 12-week supervised aerobic training regimen.

A total of 120 healthy home residents and older subjects with an age range of 65 to 95 years were enrolled to participate in this study. Only, 60 subjects who met the inclusion criteria were included in this study.

The participants were categorized into two groups, specifically the control group (consisting of 30 individuals) and the exercise group (also comprising 30 individuals), based on their participation in an exercise program. Assessments of cognitive function, leisure-time physical activity (LTPA), and apoptotic-related markers such as Bcl-2, p53, and Cytochrome c were conducted both before and after a 12-week aerobic exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* home resident older
* healthy individuals
* the participants were aged between 65 and 95

Exclusion Criteria:

* Participants with Any physical impairments or conditions such as endocrine, immune, or psychiatric disorders
* participants with eating disorders
* participants' use of any glucocorticoid medications, which might impact the assessment of apoptotic and cognitive functions.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12-25 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of body weight as anthropometric measurements | 3 month
  the impact of exercise training program on body weight was identified pre and post exercise period. Weight measurements in kilograms from all participants were estimated by employing a standardized approach, utilizing a tape measure and a calibrated Salter Electronic Scale (Digital Pearson Scale; ADAM Equipment Inc., Columbia, MD, USA). The calculated weights were used to estimate BMI of each recpective participant.
Assessment of body height as anthropometric measurements | 3 month
  the impact of exercise training program on body height was identified pre and post exercise period. A standardized approach, utilizing a tape measure and a calibrated Salter Electronic Scale (Digital Pearson Scale; ADAM Equipment Inc., Columbia, MD, USA) were used to estimate body height of each participants. The values of body height in meters were used in combination with body weight to perform BMI of its respective participant.
Assessment of BMI as as anthropometric measurements | 3 month
  Assessment of body mass index ( BMI in kg/m^2)as anthropometric measurements In this test, BMI from body weight and height measurements for each participant were estimated before and after exercise training interventions by using a bioelectrical impedance analysis (BIA) based body composition analyzer (TBF 105, Tanita Corporation, Tokyo, Japan)

SECONDARY OUTCOMES:
Assessment of cognitive abilities | 3 month
  the cognitive capabilities of the elderly participants prior and post structured aerobic exercise program using the Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) battery.The LOTCA comprises seven primary domains, each further subdivided into 26 subtests. Scoring for each subtest was carried out utilizing either a four- or five-point Likert scale. The overall LOTCA score was obtained by summing the scores from all subtests. Scores on the test range from a minimum of 27 to a maximum of 123, where a higher score signifies superior cognitive function.
Assessment of serum Bcl-2 as apoptotic-related protein | 3 month
  in this outcome measure, ELISA kits specifically designed for Bcl-2 (Cat# QIA23, Oncogene Research Products, Germany). The levels of serum Bcl-2 (µg/ml) were identified in all participants of control and exercised groups, pre- and post exercie training for 12 weeks
Assessment of serum cytochrome c as apoptotic-related protein | 3 month
  Serum cytochrome c (ng /ml) was estimated in the serum of all participant's by using cytochrome c (Zymed ELISA Kit, Cat. No. 99-0040). The results were measured by immunoassay analysis using ELISA reader
Assessment of serum p53 (pg/ml) as apoptotic-related protein | 3 month
  The quantification of p53 (pg/ml) concentration in the serum of all participants before and after exercise training was determined utilizing a single-step enzyme-immunoassay ELISA kit (Catalog Number 11 828 789 001; Roche Diagnostics GmbH, Roche Applied Science, Germany) based on photometric methods.